CLINICAL TRIAL: NCT00126152
Title: Targeted Injury Prevention Program: Preventing Falls Among Older Adults
Brief Title: Senior Falls Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State, Department of Health (Other Government)
Collaborators: NorthWest Orthopaedic Institute (Other); Spokane Regional Health District (Unknown); University of Washington (Other); Senior Services of Seattle/King County (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: U17/CCU022310
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2005-08-02 (Estimated); Status verified 2005-07

CONDITIONS: Falls Among Older Adults
Keywords: Falls; Exercise; Fall Risk Factors; Older Adults
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Educational Status

INTERVENTIONS:
Behavioral: Exercise, education and medical management

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a best practice model for senior falls prevention when implemented in a community setting.

DETAILED DESCRIPTION:
This study will measure differences in the incidence of falls and fall risk factors among subjects assigned to an intervention group and a control group. Subjects in the intervention group will receive a multi-faceted intervention based on best practices. Subjects in the control group will receive written fall prevention education materials. Fall monitoring will be conducted for subjects in both groups.

Specific components of the intervention will include:

* an individual fall risk assessment;
* exercise with balance and strength training;
* education on how to reduce falls and fall risk factors; and
* recommendations for medical care management of identified fall risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older;
* Live in the community in a house, apartment, or retirement center;
* Able to speak and understand English;
* Able to walk without the physical assistance of another person (using an assistive device, such as a cane or walker, is ok);
* Able to participate in a falls prevention program for 12 months;
* Able to participate in exercise classes that meet 3 times per week for a minimum of 6 months.
* Able to provide their own transportation and be a year-round resident;
* Have a health care provider that they had seen within the past three years;
* Able to see and hear another person from a distance of 10 to 12 feet.
* Able to complete a 10-foot Timed Up and Go Test in < 30 seconds.
* Able to complete the Pfeiffer Short Portable Mental Status Questionnaire with fewer than 5 errors.

Exclusion Criteria:

* Participated in regular, moderate exercise during the past 3 months (Regular exercise means physical activity that is done 30 minutes or longer, 3 or more times a week. Moderate exercise includes any physical activity that makes the heart beat faster or makes a person breathe harder or sweat, such as brisk walking, active gardening, or climbing stairs.)
* Has Parkinson disease or multiple sclerosis;
* Is under doctor's orders to restrict activity level.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 453
Dates: Start 2003-09; Study Completion 2005-05

PRIMARY OUTCOMES:
Change in the incidence of falls, reported once a month over a one year follow-up period.

SECONDARY OUTCOMES:
Changes in lower body strength, balance and mobility measured at baseline and repeated at the end of a one year follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Mary K LeMier, MPH, Principal Investigator — Washingon State Department of Health, Injury & Violence Prevention Program; Ilene F Silver, MPH, Principal Investigator — Washington State Department of Health, Injury & Violence Prevention Program
Locations (2):
- United States (2):
  - Spokane Regional Health District, Spokane, Washington
  - Northwest Orthopaedic Institute, Tacoma, Washington